CLINICAL TRIAL: NCT01053936
Title: A Multi-Center, Open-Label, Randomized, Parallel Group, Dose-Ranging, Pharmacodynamic Phase II Trial to Determine the Effects of Bardoxolone Methyl (RTA 402, Amorphous Dispersion) on eGFR in Patients With Type 2 Diabetes and Chronic Kidney Disease (eGFR 15-45 mL/Min/1.73m2)
Brief Title: Phase II Pharmacodynamic Trial to Determine the Effects of Bardoxolone Methyl on eGFR in Patients With Type 2 Diabetes and Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTA 402-C-0902
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2
Keywords: Chronic Kidney Disease; Type 2 diabetes; Diabetic Nephropathy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — bardoxolone methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Bardoxolone methyl: 5 mg (Experimental)
  Interventions: Drug: Bardoxolone methyl (amorphous dispersion)
- Bardoxolone methyl: 10 mg (Experimental)
  Interventions: Drug: Bardoxolone methyl (amorphous dispersion)
- Bardoxolone methyl: 15 mg (Experimental)
  Interventions: Drug: Bardoxolone methyl (amorphous dispersion)
- Bardoxolone methyl: 30 mg (Experimental)
  Interventions: Drug: Bardoxolone methyl (amorphous dispersion)
- Bardoxolone methyl: 2.5 mg (Experimental)
  Interventions: Drug: Bardoxolone methyl (amorphous dispersion)

INTERVENTIONS:
Drug: Bardoxolone methyl (amorphous dispersion) — Oral, once daily

SUMMARY:
This study assesses the effects of a new formulation of bardoxolone methyl on eGFR in Patients with Chronic Kidney Disease and Type 2 Diabetes.

DETAILED DESCRIPTION:
Bardoxolone methyl (RTA 402) is an Antioxidant Inflammation Modulator (AIM) that is undergoing clinical testing in chronic kidney disease (CKD). Bardoxolone methyl and other AIMs inhibit immune-mediated inflammation by restoring redox homeostasis in inflamed tissues through the induction of the cytoprotective transcription factor Nrf2. In the diabetic population, adipocytes produce cytokines and mobilize free fatty acids which induce insulin resistance. Resultant hyperglycemia and increased cytokine production induces reactive oxygen and nitrogen species which in turn induce vascular inflammation and endothelial dysfunction. These stimuli cause further activation of NF-kB, promoting inflammation, mesangial cell contraction, mesangial expansion and endothelial dysfunction, the end result of which is decreased renal function. By inducing Nrf2 and suppressing redox-driven inflammation, we hypothesize that inflammation and resultant adverse renal functional changes in patients with chronic kidney disease resulting from diabetes can be suppressed.

In a Phase IIa open label study of patients with CKD and type 2 diabetes, treatment with bardoxolone methyl for 28 days resulted in significant improvements in renal function, including increases in eGFR, and decreases in serum creatinine, cystatin C, BUN, phosphorus, uric acid, creatinine clearance, and angiotensin II; improvements in glycemic control as assessed by hemoglobin A1c; and improvements in markers of endothelial dysfunction and systemic inflammation, such as circulating endothelial cells and adiponectin. These data are consistent with the hypothesis that bardoxolone methyl improves renal function through suppression of renovascular oxidative stress and inflammation.

A new formulation of bardoxolone methyl has been developed, which is the same chemical entity but manufactured to contain an amorphous dispersion rather than a crystalline solid state. The new amorphous dispersion formulation of bardoxolone methyl has been shown to be more orally bioavailable in non-human primates. The purpose of this study is to determine the appropriate dose of the new bardoxolone methyl formulation to use in future clinical studies by determining the dose response relationship on eGFR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a history of type 2 diabetes; diagnosis of type 2 diabetes should have been made at >30 years of age (if diabetes developed at a younger age, C-peptide level may be obtained to confirm diagnosis);
2. Patients must be at least 18 years of age;
3. The average of 2 eGFR values collected during screening must be within 15 - 45 mL /min/1.73m2 inclusive.
4. Patients must be receiving an angiotensin converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB) for at least 8 weeks prior to screening, where the dose of the ACE inhibitor or the ARB is considered appropriate for that patient, and the patient has been stable and maintained on that dose for at least 8 weeks prior to randomization (Day 1). No change in ACE or ARB therapy should be anticipated or planned for the period of the study.
5. Male and female patients must agree to use effective contraception during the entire study period and for at least 2 months after the last dose of study drug, unless documentation of infertility exists
6. Women of child-bearing potential must have a negative serum pregnancy test result at screening and a confirmed negative urine pregnancy test result prior to administration of the first dose of study medication;
7. Patient is willing and able to cooperate with all aspects of the protocol;
8. Patient is willing and able to give written informed consent for study participation

Exclusion Criteria:

1. Any patient with Type 1 (insulin-dependent; juvenile onset) diabetes; or any history of diabetic ketoacidosis;
2. Any patient with known non-diabetic renal disease, family history of a hereditary form of kidney disease, or patients with a history of a renal transplant.
3. Any patient with clinical or renal biopsy evidence of any non-diabetic renal disease other than nephro-sclerosis;
4. Any patient with blood pressure (BP) that is unable to be controlled to a systolic pressure (SeSBP) <160 mmHg and a diastolic pressure (SeDBP) of <90 mmHg. BP will be determined by the average of 3 readings, taken after being seated for at least 5-minutes. BP must be within this range taken at 2 separate time-points at least 4 days apart during the screening period;
5. Any patient with Hemoglobin A1c level >10% collected at screening;
6. Any patient with cardiovascular disease as follows:

   1. Unstable angina pectoris within 3 months before study randomization;
   2. Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 3 months before study randomization;
   3. Transient ischemic attack within 3 months before study randomization;
   4. Cerebrovascular accident within 3 months before study randomization;
   5. Obstructive valvular heart disease or hypertrophic cardiomyopathy;
   6. 2nd degree or 3rd degree atrioventricular block not successfully treated with a pacemaker;
   7. Current diagnosis of Class III or IV congestive heart failure ;
7. Any patient with QTc Fredericia interval > 450 milliseconds as determined by the average of values reported by a central reader from 3 ECGs taken at the Screening Visit.
8. Any patient with need for chronic (>2 weeks) immunosuppressive therapy, including corticosteroids (excluding intra-articular injections inhaled or nasal steroids) within 3 months prior to randomization;
9. Any patient who requires more than occasional (once or twice weekly) use of non-steroidal anti-inflammatory agents (NSAIDS);
10. Any patient who requires a change or dose adjustment in any of the following medications: ACE inhibitors and ARBs within 8 weeks; other anti-hypertensive, and other anti-diabetic medications within 6 weeks prior to study randomization;
11. Any patient who is unable or unwilling to discontinue the following medications throughout the study period: Niacin® (nicotinic acid), Niaspan® (nicotinic acid), Niacor® (nicotinic acid), Nicolar® (nicotinic acid),Nicobid® (nicotinic acid), Nydrazid® (isoniazid), Dantrium® (dantrolene), Normodyne® (labetalol), Trandate® (labetalol), Cylert® (pemoline), Tradon® (pemoline), PemADD® (pemoline), Felbatol® (felbamate), Zyflo® (zileuton),Tasmar® (tolcapone), or Tricor® (fenofibrate), Antaram® (fenofibrate), Triglide® (fenofibrate), Lofibra® (fenofibrate), Lipidil Micro® (fenofibrate), Lipidil Supra® (fenofibrate); including fenofibrate derivatives e.g. Lopid® (gemfibrozil) and Atromid-S® (clofibrate) . Patient must discontinue the aforementioned medications for a minimum of two weeks prior to randomization. Patients may continue use of multi-vitamins (e.g., Centrum) ®, which have a maximum total daily consumption of <= 50 mg of nicotinic acid (Niacin®);
12. Any patient with evidence of hepatic or biliary dysfunction including levels of total bilirubin >1.0 mg/dL (>17 micromole/L), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > upper limit of normal (ULN), or alkaline phosphatase >2.0 times the ULN on ANY screening laboratory test result;
13. If a patient provides a history of hepatitis B or C but has normal liver enzyme levels, the investigator should perform a serologic hepatitis screen and call the Medical Monitor to discuss patient eligibility. Patients with a history of hepatitis A that is resolved and who do not demonstrate any liver enzyme level elevation are eligible for protocol randomization;
14. Any female patient who is pregnant, nursing or planning a pregnancy;
15. Any patient with known hypersensitivity to any component of the study drug;
16. Any patient who has undergone diagnostic or intervention procedure requiring a contrast agent within the last 30 days prior to study randomization;
17. Patient with a current history of drug or alcohol abuse as per the Investigator's assessment;
18. Any patient with a history of neoplastic disease (except basal or squamous cell carcinoma of the skin) within 5 years prior to study randomization;
19. Any patient who has had dialysis within 3 months before randomization and/or have not maintained a stable level of kidney function within 3 months of randomization per Investigator assessment;
20. Any patient who has any concurrent clinical conditions that in the judgment of the investigator could either potentially pose a health risk to the patient while involved in the study or could potentially influence the study outcome;
21. Any patient who has participated in another clinical study involving investigational or marketed products within 30 days prior to randomization or would concomitantly participate in such a study, or any patient who has received bardoxolone methyl in any form;
22. Any patient who is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-01-31 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2011-02-28 (Actual)

PRIMARY OUTCOMES:
To assess a trend in mean change from baseline to Day 29 in eGFR (as estimated by the 4-component MDRD formula) with increasing doses of bardoxolone methyl (amorphous dispersion) in patients with Type 2 diabetes and CKD (eGFR 15-45 mL/min/1.73m2). | 29 Days

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of bardoxolone methyl (amorphous dispersion) after 28 and 84 days of administration. | 85 days
To assess a trend in mean change from baseline to Day 85 in eGFR (as estimated by the 4-component MDRD formula with increasing doses of bardoxolone methyl (amorphous dispersion) in patients with Type 2 diabetes and CKD (eGFR 15-45 mL/min/1.73m2) | 85 days

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Montgomery, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - La Mesa, California
  - Riverside, California
  - San Dimas, California
  - Washington D.C., District of Columbia
  - Brandon, Florida
  - Port Charlotte, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Canton, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Brooklyn Center, Minnesota
  - Morehead City, North Carolina
  - Winston-Salem, North Carolina
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Chattanooga, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Greenville, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Federal Way, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/